CLINICAL TRIAL: NCT03279497
Title: Health Game Intervention to Promote the Physical Activity of Early Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Anni Pakarinen, Doctoral candidate, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MoveF2017
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Physical Activity; Health Behavior
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health game (Experimental): Health game intervention consists of 20 minutes guided training session with the mobile health game at school and 4 weeks free usage of the game via own smart phone during free time. Smart phones are tracking the actual physical activity (steps) of the participants via activity sensors and the tracked steps work as In-App Currency enabling the participants to play the game and proceed in it.
  Interventions: Behavioral: Health game
- Sport and fitness application (Sham Comparator): Sport and fitness application intervention consists of 20 minutes guided training session with the app at school and 4 weeks free usage of the app via own smart phone during free time. Sport and fitness application, when turned on, tracks the physical activity (running, cycling and every-day training) of the participant.
  Interventions: Behavioral: Sport and fitness application

INTERVENTIONS:
Behavioral: Health game — Participants allocated to the Health game intervention group get to use the health game during the four week intervention period and participants are allowed to use it on their free time.
  Arms: Health game
Behavioral: Sport and fitness application — Participants allocated to the Sport and fitness application intervention group get to use the sport and fitness application during the four week intervention period and participants are allowed to use it on their free time.
  Arms: Sport and fitness application

SUMMARY:
The study evaluates the effectiveness of the game-intervention in promotion of physical activity self-efficacy and physical activity behavior among early adolescents (10-13 year olds). Half of the study participants will receive the game-intervention and half of the study participants will receive a commercially available sport and fitness application for running, cycling and every-day training.

DETAILED DESCRIPTION:
The study evaluates the effectiveness of the game-intervention in promotion of physical activity self-efficacy and physical activity behavior among early 10 to 13 years old adolescents. Participants allocated to the Health game intervention group will use a game called Movenator, during a four week intervention and participants allocated to the Sport and fitness-intervention group will use a commercially available Sport and fitness application for running, cycling and every-day training, during a four week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Goes to school at 4th, 5th or 6th grade
* Understands and can communicate either in Finnish
* Has daily access to a smart phone (Android) during free time

Exclusion Criteria:

* Physical activity impairments

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical activity behavior | at baseline during one week period and at 4 weeks during one week period
  Physical activity behavior is tracked with Actigraph wGT3X-BT accelerometer during one week period

SECONDARY OUTCOMES:
Change in Physical activity self-efficacy | At baseline and at 4 weeks
  Measured with Physical Activity Self-Efficacy Scale (PASES), a 8-item 5-point Likert-scale.
Actual use of the intervention | During the four week intervention
  Actual use of the intervention is tracked with log files
Usability of the intervention | At 4 weeks
  Measured with System Usability Scale (SUS), a 10-item 5-point Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Anni Pakarinen, MHSc, Principal Investigator — University of Turku
Locations (1):
- Primary schools (n=2), Turku, Southwest Finland, Finland